CLINICAL TRIAL: NCT00746967
Title: An Open-Label, Multi-Center Extension Study To Evaluate The Safety, Toleration And Sustained Efficacy Of Oral Sildenafil Administered To Women Who Have Been Diagnosed With Female Sexual Arousal Disorder
Brief Title: An Open-Label, Extension Study Evaluating the Safety, Toleration, and Efficacy of Sildenafil in Women With Sexual Arousal Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481133
Record Dates: First submitted 2008-03-31; First posted 2008-09-04 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Sexual Dysfunctions, Psychological; Sexual Arousal Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Sildenafil Citrate

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: sildenafil

INTERVENTIONS:
Drug: sildenafil — sildenafil 50 mg (starting dose) tablet by mouth taken as needed 1 hour before anticipated sexual activity; the dose could be increased to 100 mg or decreased to 25 mg; the duration of therapy in this open-label study was 52 weeks

SUMMARY:
The purpose of this study is to evaluate the safety and toleration of oral sildenafil administered as required by women with Female Sexual Arousal Disorder (FSAD) who successfully complete one of the following Pfizer-sponsored, 12-week, double-blinded clinical trials: A1481082 or A1481123. Addition of this 52-week open-label extension will increase the total duration of sildenafil exposure to 64 weeks. Sustained efficacy will also be evaluated after 3 and 6 months of open-label therapy.

ELIGIBILITY:
Inclusion Criteria:

* Included were subjects who completed Pfizer study A1481082 or A1481123 without a major protocol violation and with all treatment-related adverse events resolved prior to crossover into the open-label study.
* For subjects receiving hormone replacement therapy and/or selective serotonin reuptake inhibitor treatment, dosage of these must be stable at the start of this extension study and remain stable throughout.
* Subjects should continue to maintain a stable sexual relationship throughout the study.

Exclusion Criteria:

* Excluded were subjects who experienced either treatment-related serious adverse events or significant treatment-related laboratory abnormalities in the previous study, and subjects who misused study medication and/or failed to adequately account for study medication in the previous study, or who were non-compliant with visits.
* Also excluded were subjects who were currently prescribed and/or taking nitrates or nitric oxide donors in any form (oral, sublingual, buccal, transdermal, inhalational or aerosols).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2003-01; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Safety/toleration of oral sildenafil. | Continuous

SECONDARY OUTCOMES:
The score for each of the individual questions 3,5 and 9 on the SQoL-F | Week 14 and Week 26
The total satisfaction score on the Inventory of Treatment Satisfaction (ITS-modified EDITS) | Week 14 and Week 26
The score for each of the individual questions 3,5,6 and 7 on the ITS-modified EDITS | Week 14 and Week 26
The Arousal-lubrication Domain from the SFQ. The score for this domain is the sum of scores from Questions 11 and 12 from the SFQ | Week 14 and Week 26
The Arousal-sensation Domain from the SFQ. The score for this domain is sum of scores from Questions 7,8,9 and 10 from the SFQ. | Week 14 and Week 26
The total Quality of Life score on the Sexual Quality of Life (SQoL-F) | Week 14 and Week 26
The Desire domain from the SFQ. Specifically, the sum of scores from questions 1,2,3,4,15 and 28 (frequency of pleasurable thoughts, wanted to be touched, wanted sex, initiated sex, had sex with penetration, looked forward to sex, respectively). | Week 14 and Week 26
Question 16 from the SFQ at Weeks 14 and 26 (enjoyment of penetration and intercourse). | Week 14 and Week 26
The Orgasm domain from the SFQ. The score for this domain is the sum of scores from questions 24,25 and 26 (orgasm frequency, level of pleasure and ease in achieving, respectively). | Week 14 and Week 26
The individual questions of the Orgasm domain. | Week 14 and Week 26
SFQ Question 27 (confidence as sexual partner). | Week 14 and Week 26
SFQ Question 29 (disappointment with response). | Week 14 and Week 26
Global Efficacy Question (SFQ Question 34, satisfaction with whole of sexual life) | Week 14 and Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- United States (71):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Anchorage, Alaska
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Jonesboro, Arkansas
  - Pfizer Investigational Site, Albany, California
  - Pfizer Investigational Site, Berkeley, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Burbank, California
  - Pfizer Investigational Site, Fair Oaks, California
  - Pfizer Investigational Site, Hermosa Beach, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, New London, Connecticut
  - Pfizer Investigational Site, Waterbury, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Brooksville, Florida
  - Pfizer Investigational Site, Jensen Beach, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Leawood, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Florence, Kentucky
  - Pfizer Investigational Site, Metairie, Louisiana
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Creve Coeur, Missouri
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, North Las Vegas, Nevada
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, White Plains, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Reading, Pennsylvania
  - Pfizer Investigational Site, Temple, Pennsylvania
  - Pfizer Investigational Site, West Reading, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Sandy City, Utah
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, Cheyenne, Wyoming

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481133&StudyName=An%20Open-Label%2C%20Extension%20Study%20Evaluating%20the%20Safety%2C%20Toleration%2C%20and%20Efficacy%20of%20Sildenafil%20in%20Women%20With%20Sexual%20Arousal%20Disorder.%0A